CLINICAL TRIAL: NCT00000245
Title: Evaluation of a Desipramine Ceiling in Cocaine Abuse
Brief Title: Evaluation of a Desipramine Ceiling in Cocaine Abuse - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Friends Research Institute, Inc. (Other)
Purpose: Treatment
Other Study IDs: NIDA-08082-1; R01-08082-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Desipramine

INTERVENTIONS:
Drug: Desipramine

SUMMARY:
The purpose of this study is to confirm whether a blood level ""ceiling"" exists on desipramine effect in cocaine abuse.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1994-05; Study Completion 2001-12

PRIMARY OUTCOMES:
Craving
Retention
Cocaine use
Depression
Anxiety
Mood indicators

CONTACTS AND LOCATIONS:
Overall Officials: Frank Gawin, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States